CLINICAL TRIAL: NCT06395337
Title: A Phase I/II Study to Evaluate the Safety and Feasibility of Multimodal Imaging Using a Dual-labeled Anti-CEA Antibody in Patients With Rectal or Pancreatic Cancer
Brief Title: Multimodal Imaging in Rectal Cancer & Pancreatic Cancer
Acronym: MIRCA & MIPAC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: Leiden University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ORG-100023234
Record Dates: First submitted 2024-04-09; First posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2023-07

CONDITIONS: Rectal Cancer; Pancreatic Cancer
MeSH Terms: conditions — Rectal Neoplasms; Pancreatic Neoplasms | interventions — Mastectomy, Segmental

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intraoperative multi-modality imaging (Experimental): Patients receive a single intravenous dose of [111In]In-DOTA-ANTI-CEA antibody. At day 4 or 5 after antibody injection a SPECT/CT scan will be acquired. At day 6 or 7 standard of care cytoreductive surgery will be performed. This will be extended with the use of dual-modality imaging.
  Interventions: Drug: [111In]In-DOTA-ANTI-CEA antibody injection; Radiation: SPECT/CT scan; Procedure: Resection surgery

INTERVENTIONS:
Drug: [111In]In-DOTA-ANTI-CEA antibody injection — tracer injection
Radiation: SPECT/CT scan — abdominal and thoracic SPECT/CT scan
Procedure: Resection surgery — oncological resection surgery will be performed extended with the use of dual-modality imaging.

SUMMARY:
Most digestive cancers show (over)expression of the tumour marker carcinoembryonic antigen (CEA). Therefore, interest in CEA-targeting tracers has increased over the past years. CEA-targeting tracers can be used for preoperative, intra-operative and postoperative imaging purposes. This study focusses on both preoperative and intraoperative multimodal imaging and image-guided surgery in patients with rectal cancer or pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of rectal cancer where a (beyond) TME resection is planned for OR Clinical suspicion of PDAC
* Scheduled for surgical resection
* Age over 18 years
* Signed informed consent

Exclusion Criteria:

* Any medical condition present that in the opinion of the investigator will affect patients' clinical status
* Administration of a radionuclide within 10 physical half-lives prior to study enrollment
* Pregnancy or lactation
* Known CEA negative tumor: If a patient had a primary tumor which did not express CEA determined immunohistochemically on the resection specimen of a prior operation or biopsy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-05-02 (Estimated); Primary Completion 2025-05-02 (Estimated); Study Completion 2025-06-02 (Estimated)

PRIMARY OUTCOMES:
Safety of dual-labeled antibody as assessed by the number of participants with grade 3 or 4 Adverse Events according to CTCAE v4.0 | 30 days
  Safety of dual-labeled antibody injection as assessed by the number of participants with grade 3 or 4 Adverse Events according to CTCAE v4.0

SECONDARY OUTCOMES:
Intensity of fluorescence | 7 days
  To assess the intensity of fluorescence in malignant and non-malignant tissue, using quantifiable images
Intensity of radiosignal | 7 days
  To assess the intensity of the radiosignal in malignant and non-malignant tissue, using radioactive measuring device.
Concordance between CEA and tracer | 7 days
  To assess the concordance between localization of the [111In]In-ANTI-CEA and CEA expression in rectal or pancreatic cancer and non-malignant tissue, by analyzing pathologic tissue for tracer activity and CEA presentation
Blood levels of the dual-labeled antibody | 30, 60, 120, 180 minutes
  To determine blood concentrations at several time points in patients to assess the pharmacokinetics of the tracer.
Biodistribution | 7 days
  To determine the whole body biodistribution of the tracer over time by quantified SPECT/CT imaging at 2 timepoints.

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Leiden University Medical Center, Leiden
  - Radboudumc, Nijmegen